CLINICAL TRIAL: NCT02660879
Title: The Effect of Video Education on Improving Inhaler Use Technique
Brief Title: The Effect of Video Education on Inhaler Use Technique
Acronym: InhalerEdu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Romil Fenil Shah (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor-Investigator, Romil Fenil Shah, Medical Student, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00087922
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Nebulizers and Vaporizers; Patient Education; E Learning
Keywords: Education; Inhaler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Written Education (Placebo Comparator): These patients were video taped before they had any inhaler education using their own inhalers. They were then given written educational materials, and given 5 minutes to read these materials. They were then re-taped for their inhaler technique.
  Interventions: Other: Written Document Educational Resource
- Online Video Education (Experimental): These patients were video taped before they had any inhaler education using their own inhalers. They were then given online video education located at use-inhalers.com, and were asked to complete the education (took on average 5 minutes). They were then re-taped for their inhaler technique.
  Interventions: Other: Online Video Education

INTERVENTIONS:
Other: Written Document Educational Resource — A 2 page document with pictures discussing how to use an inhaler properly.
  Arms: Written Education
Other: Online Video Education — Education which included step-by-step instruction on how to use their inhalers correctly as well as a webcam element that allowed users to see themselves practice their inhalers along with actors on screen.
  Arms: Online Video Education

SUMMARY:
The investigators looked at the effect that video instruction located at www.useinhalers.com would have on improving inhaler technique at a hospital in Guayaquil, Ecuador. The investigators compared this video instruction to written Spanish inhaler education. The investigators video taped participants before and after the intervention, and graded their technique on a pre-defined rubric.

ELIGIBILITY:
Inclusion Criteria:

* Clinically-stable outpatient adults (≥18 years) with Asthma or Chronic Obstructive Pulmonary Disease (COPD) with history of at least one exacerbation in last 1 year
* Clinical diagnoses of asthma or COPD

Exclusion Criteria:

* Patients with language barrier (unable to understand and communicate in either English or Spanish)
* Cognitive or physical dysfunction that, in the investigator's opinion, would interfere with completion of the study
* Significant co-morbidity that can confound asthma symptoms - e.g. Congestive Heart Failure, current smoker, uncontrolled Gastroesophageal Reflux Disease, neuromuscular disease, chest wall deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Inhaler Technique Defined by 11 point rubric which details steps and techniques necessary for proper inhaler use | Videos taken before educational interventions and directly after the 5-10 minutes allotted for the educational intervention. Videos will be assessed in the following months after using the 11 point rubric.

REFERENCES:
- [Background] http://www.cdc.gov/VitalSigns/Asthma (accessed: 28 July 2012)
- [Background] Press VG, Arora VM, Shah LM, Lewis SL, Ivy K, Charbeneau J, Badlani S, Nareckas E, Mazurek A, Krishnan JA. Misuse of respiratory inhalers in hospitalized patients with asthma or COPD. J Gen Intern Med. 2011 Jun;26(6):635-42. doi: 10.1007/s11606-010-1624-2. Epub 2011 Jan 20. PMID 21249463
- [Background] Hagmolen of ten Have W, van de Berg NJ, Bindels PJ, van Aalderen WM, van der Palen J. Assessment of inhalation technique in children in general practice: increased risk of incorrect performance with new device. J Asthma. 2008 Jan-Feb;45(1):67-71. doi: 10.1080/02770900701815834. PMID 18259998
- [Background] Fink JB, Rubin BK. Problems with inhaler use: a call for improved clinician and patient education. Respir Care. 2005 Oct;50(10):1360-74; discussion 1374-5. PMID 16185371
- [Background] Al-Jahdali H, Ahmed A, Al-Harbi A, Khan M, Baharoon S, Bin Salih S, Halwani R, Al-Muhsen S. Improper inhaler technique is associated with poor asthma control and frequent emergency department visits. Allergy Asthma Clin Immunol. 2013 Mar 6;9(1):8. doi: 10.1186/1710-1492-9-8. PMID 23510684
- [Background] Cavender A, Alban M. Compulsory medical service in Ecuador: the physician's perspective. Soc Sci Med. 1998 Dec;47(12):1937-46. doi: 10.1016/s0277-9536(98)00335-9. PMID 10075237
- [Derived] Shah RF, Gupta RM. Video instruction is more effective than written instruction in improving inhaler technique. Pulm Pharmacol Ther. 2017 Oct;46:16-19. doi: 10.1016/j.pupt.2017.08.005. Epub 2017 Aug 7. PMID 28797611